CLINICAL TRIAL: NCT03527992
Title: Automated Oxygen Administration in Patients With Hypoxemic Pneumonia and Pleuropneumonia
Acronym: OPPAÎ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/17/0404; 2017-A03642-51 (Other: ID-RCB)
Record Dates: First submitted 2018-03-08; First posted 2018-05-17 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Pneumonia; Pneumonia, Ventilator-Associated; Length of Stay
Keywords: Randomized Therapeutic trial; Hypoxemic pneumonia; Automated oxygen therapy; Length of stay; medico-economic cost
MeSH Terms: conditions — Pneumonia; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automated oxygen therapy (Other): An automated oxygen therapy is a system that allows administration of oxygen with a flow that is automatically adjusted to the patient's saturation, which is continuously monitored. Patients will receive O2 automated intervention.
  Interventions: Device: O2 automated
- Standard Oxygen therapy (Other): Patients will receive O2 standard therapy
  Interventions: Device: O2 standard

INTERVENTIONS:
Device: O2 automated — In the "O2 automated" group, patients benefit from oxygen therapy via the "FreeO2" device. The O2 saturation target is set by the clinician on the device. Saturation is continuously sensed by an oximeter and the oxygen flow is automatically adjusted. The clinician has access to instantaneous values and trends of O2 and SpO2 flow rates.
  Arms: Automated oxygen therapy
Device: O2 standard — In the "O2 standard" group, patients benefit from oxygen therapy with nasal goggles or a high concentration mask. Saturation is continuously captured by an oximeter. The flow rate of oxygen, evaluated in L/min, is adapted according to local protocols (every 8 hours in conventional hospital services, continuous in intensive care
  Arms: Standard Oxygen therapy

SUMMARY:
Hypoxemic pneumonia is a major cause of hospitalization in Pulmonology. The patient's dependency on oxygen prevents early discharge from the hospital. An automated oxygen therapy is a system that allows administration of oxygen with a flow that is automatically adjusted to the patient's saturation, which is continuously monitored. This system has proven to be particularly effective with chronic obstructive pulmonary disease (COPD) patients, by decreasing the time spent in hypoxia and hyperoxia, and by accelerating the weaning of oxygen. Our hypothesis is that automated oxygen therapy leads to a diminution on the length of hospital stay.

DETAILED DESCRIPTION:
Prolonged hospitalization has many consequences, including loss of autonomy and nosocomial infection. Moreover, these complications themselves lead to an extension of the length of stay. This has an impact on the cost of care: several studies have shown that hospitalization is the most costly factor in the management of pneumonia, and that even a small amount of hospital stay, led to significant financial savings. Automated oxygen therapy is a device that automatically adjusts with the saturation the amount of oxygen administered. Investigator hypothesis is that automated oxygen therapy could shorten the length of stay of patients hospitalized for hypoxemic pneumonia. One group of patients will receive the automated oxygen therapy and the other group will receive the standard Oxygen therapy. The investigator will compare in each group the average length of stay, the duration of oxygen therapy, the time spent outside of the target saturation, the cost on the medical-economic level and the patient's experience.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Patient living at home or in an institution
* Patient hospitalized for less than 48 hours
* Pneumonia defined (according to the 2006 French-speaking infectious pneumology society (SPILF) criteria) by:

  * respiratory functional symptoms (cough, sputum, dyspnea, chest pain) and
  * Hyperthermia >38,5°C or hypothermia <36°C and
  * Radiological Signs of Pneumonia
* Hypoxia : SpO2 < 94% in ambient air and/or PaO2< 60 mmHg in ambient air

Exclusion Criteria:

* Pneumonia acquired at the hospital.
* Patient hospitalized in another department more than 48 hours before admission
* Chronic respiratory failure
* Active neoplasia
* Patients undergoing oxygen therapy and / or long-term NIV
* Associated cardiac decompensation (clinical signs and / or NTproBNP> 1800ng / mL) (3
* Initial Need for high flow oxygen therapy or ventilatory support (NIV, VI)
* Difficulties expected from home support.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2018-03-09 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Length in days of hospital stay | 1 month
  measure of total days of hospitalization and intensive care

SECONDARY OUTCOMES:
Duration of oxygen therapy | 1 month
  Oxygen therapy time evaluation during hospitalization of patient
Time spent outside of the target saturation | 1 month
  Investigator want evaluate the time spent outside of the target saturation by patient, during their hospitalization,
the cost on the medical-economic level | 1 month
  investigator want evaluate the cost of hospitalization between patient in arm "Automated oxygen therapy" and patient in arm "Standard Oxygen therapy"
rate of medical complication | 1 month
  Investigator want to evaluate the rate of medical complication between patient in arm "Automated oxygen therapy" and patient in arm "Standard Oxygen therapy"
quality questionnaire of patient's life during hospitalization | 1 month
  Investigator want to evaluate the quality of life during hospitalization between patient in arm "Automated oxygen therapy" and patient in arm "Standard Oxygen therapy"

CONTACTS AND LOCATIONS:
Overall Officials: Elise Noel-Savina, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Larrey, Toulouse, France

IPD SHARING:
Plan to Share IPD: No